CLINICAL TRIAL: NCT00054938
Title: A Randomized Controlled Trial of Strategies for the Prevention of Accelerated Atherosclerosis in Systemic Lupus Erythematosus - A Pilot Study
Brief Title: Prevention of Atherosclerosis and Heart Disease in Patients With Systemic Lupus Erythematosis (SLE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Matthew H. Liang, MD, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P60 AR47782 NIAMS-077; P60AR047782 (NIH)
Record Dates: First submitted 2003-02-13; First posted 2003-02-14 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Systemic Lupus Erythematosus; Lupus
Keywords: SLE; Accelerated Atherosclerosis; Cholesterol
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Pravastatin; Aspirin; Ramipril; Vitamin B 12; Folic Acid

INTERVENTIONS:
Drug: pravastatin
Drug: aspirin
Drug: ramipril
Drug: Vitamins: B6, B12, and folate
Behavioral: heart health educational program

SUMMARY:
The purpose of this study is to find the best way to prevent heart disease and stroke in people with lupus (systemic lupus erythematosis, or SLE). The study will evaluate the effectiveness of medication and a phone-based education program in controlling four risk factors for heart disease: smoking, obesity, high blood pressure, and inactivity. The study will also test the safety of commonly used heart medications in people with lupus.

DETAILED DESCRIPTION:
People with SLE are at much higher risk for mortality due to atherosclerotic vascular disease (ASVD). Available data suggest that the usual mechanics of and risk factors for atherosclerosis are enhanced by factors such as corticosteroid use and SLE itself. This study will evaluate a medication and education program designed to prevent ASVD complications (primary prevention) or their recurrence (secondary prevention). The study will also measure the compliance and retention rate for the prevention program over 4 years.

Participants in this study will be randomized to receive either preventive heart disease medications or placebo. Participants in the medication arm will receive pravastatin alone or in combination with the following: aspirin, ramipril, or a combination of vitamins B6, B12, and folate. All participants in this study will receive basic education on how to optimize their heart health. Educational material will be sent to the patients as well as to support persons whom they have named. One group will receive tailored education based on a particular risk factor. Participants will have three study visits and follow-up telephone visits four times a year. Study visits will include a medical history and basic laboratory blood tests. Participants with documented high blood pressure will receive a home monitoring unit and be asked to monitor their blood pressure. Participants will be followed for 2 to 4 years.

ELIGIBILITY:
Inclusion Criteria

* SLE as defined by the 1997 American College of Rheumatology criteria
* Acceptable methods of contraception

Exclusion Criteria

* Participation in another experimental protocol for ASVD prevention
* Heavy alcohol consumption ( >= 3 drinks/day)
* Aspirin intolerance
* Certain medications, including coumadin, ACE inhibitors, potassium supplements, potassium sparing diuretics, cyclosporine, and lithium
* Peptic ulcer disease within 6 months prior to study entry
* History of an intracranial bleed or brain tumor
* Bleeding diathesis
* History of allergy or sensitivity to ACE inhibitors
* Uncontrolled high blood pressure (180 mm Hg/110 mm Hg)
* Creatinine > 2.0 mg/dl
* Renal artery stenosis
* Pregnant or breastfeeding
* Abnormal liver function tests (ALT > 2 X upper limit of normal)
* History of a muscle disease, or baseline CPK > 500U/L or 2 X upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2003-03; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew H. Liang, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, RBB Brigham Arthritis Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Liang MH, Mandl LA, Costenbader K, Fox E, Karlson E. Atherosclerotic vascular disease in systemic lupus erythematosus. J Natl Med Assoc. 2002 Sep;94(9):813-9. PMID 12392045
- [Background] Costenbader KH, Liang MH. SLE - Practical and theoretical barriers to the prevention of accelerated atherosclerosis in systemic lupus erythematosus. Arthritis Res Ther. 2003;5(4):178-9. doi: 10.1186/ar773. Epub 2003 May 23. PMID 12823848
- [Result] Costenbader KH, Karlson EW, Gall V, de Pablo P, Finckh A, Lynch M, Bermas B, Schur PH, Liang MH. Barriers to a trial of atherosclerosis prevention in systemic lupus erythematosus. Arthritis Rheum. 2005 Oct 15;53(5):718-23. doi: 10.1002/art.21441. PMID 16208639